CLINICAL TRIAL: NCT04253041
Title: Effects of Exposure to Body Positive and Fitspiration Instagram Content on Undergraduate Women's State Body Satisfaction, State Body Appreciation, and Mood
Brief Title: Social Media Effects on Lifestyle Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Socia Media and Body Image
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Control Group; Social Media

STUDY DESIGN:
Who Masked: Participant
Masking Description: To mask the true purpose of the current research and avoid biased answers related to sensitive topic such as body image and satisfaction, we will present this research as a study exploring social media's impact on lifestyle satisfaction. Visual Analogue Scales will be used to test measures of body satisfaction and appreciation, but will also include scales related to financial, social, home, and school satisfaction. At the end of this study, participants will be debriefed on the true purpose using the statement: The true purpose of this study was to examine the impacts of exposure to different Instagram images on women's body satisfaction, body appreciation, and mood. In order to understand the true effects of such without giving away the intervention, these questions were masked within a lifestyle satisfaction intervention. All of your answers will remain anonymous and will not be linked to your personal information in any way. Do you have any questions?
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): The control group will be exposed to 15 different appearance-neutral images of interior design, with a manipulation checkpoint between every other image asking participants a basic question (such as what color was most prevalent in the previous image?) regarding characteristics of the last image they were exposed to.
  Interventions: Behavioral: Effects of Instagram Exposure on Lifestyle Satisfaction
- Fitspiration (Experimental): Participants assigned to the Fitspiration condition (n=30) will be exposed to 15 different fitspiration images, with a manipulation checkpoint between every other image asking participants a basic question (such as what color was the swimsuit of the model in the previous image?) regarding characteristics of the last image they were exposed to.
  Interventions: Behavioral: Effects of Instagram Exposure on Lifestyle Satisfaction
- Body Positive (Experimental): Participants assigned to the Body Positive condition (n=30) will be exposed to 15 different body positive images, with a manipulation checkpoint between every other image asking participants a basic question (such as what color was the swimsuit of the model in the previous image?) regarding characteristics of the last image they were exposed to.
  Interventions: Behavioral: Effects of Instagram Exposure on Lifestyle Satisfaction

INTERVENTIONS:
Behavioral: Effects of Instagram Exposure on Lifestyle Satisfaction — Participants will complete initial measures of sociodemographic information, the Sociocultural Attitudes Towards Appearance Scale, The Physical Appearance Comparison Scale-Revised, and baseline measures of body appreciation, body satisfaction, and mood using online Visual Analogue Scales via Qualtrics. Female undergraduate students will be randomly assigned to one of three groups. The Fitspiration and Body Positive groups will view a series of 15 Fitspiration or Body Positive images sourced from Instagram while the control group will view 15 interior design images sourced from Instagram. After viewing images, participants will complete posttest measures of body satisfaction, body appreciation, and mood using Visual Analogue scales. Thereafter, participants will be provided with four, brief short answer questions regarding their perspective on the images observed.

SUMMARY:
From magazines to Miss America, the media has consistently contributed to the spread of sociocultural beauty standards for decades. While initial research on the effects of media on body image primarily focused on magazine and television, recent research has shifted towards exploring the effects of social media due to its rapid and constant accessibility. Current research has associated the promulgation of the thin-ideal with bulimia, dieting, supplement use, negative affect, and body dissatisfaction. Literature related to thin-ideal media (thinspiration), decreased body dissatisfaction, and negative mood is robust with a common understanding that thin-ideal media instigates increased appearance comparisons to seemingly unattainable beauty standards. Literature has also suggested that depression and anxiety have increased with the growth of social media and pressure to achieve unattainable beauty. The fit-ideal, often referred to as Fitspiration, was created as an "antidote" to thin-ideal beauty standards. However, research has found that though well intended, fitspiration content continues to promote the thin-ideal and has been associated with similarly detrimental outcomes of body dissatisfaction and negative mood. Over the last decade, body image research has shifted the focus on body disturbance to examining concepts related to positive body image. However, to date there are no known studies examining the impacts of fit-ideal content versus body positive content on women's body appreciation, body satisfaction, and state mood. The purpose of the present study is to experimentally examine the impact of exposure to body positive and fitspiration Instagram content on the body satisfaction, body appreciation, and mood of undergraduate women at Arizona State University. Participants will be 90 female undergraduate students (18-29 years old) currently attending Arizona State University. Participants will be randomly allocated to view either fitspiration, body-positive, or appearance neutral Instagram images. Dependent variables including state body appreciation, state body dissatisfaction, and state mood will be measured using Visual Analogue Scales. Trait thin-ideal internalization and trait social comparison will also be measured as moderators using the Sociocultural Attitudes Towards Appearance Questionnaire-4 and the Physical Appearance Comparison Scale-Revised. We hypothesize that viewing body positive content from Instagram will result in greater state body satisfaction, greater state body appreciation, and greater state positive mood compared to participants exposed to fitspiration and appearance neutral content. We also hypothesize that viewing fitspiration content from Instagram will result in greater state body dissatisfaction, decreased state body appreciation, and greater state negative mood compared to participants exposed to body positive and appearance neutral content. Short answer qualitative interview questions will also be included as an exploratory aim of this study where we intend to fill a gap in the literature regarding the specific aspects of each content topic that elicit the observed quantitative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Enrolled as part or full-time undergraduate students at Arizona State University
* 18-29 years old
* Access to computer and internet
* Able to read, speak, and understand English
* Willing to be randomized into one of three treatment groups

Exclusion Criteria:

* History of a clinical diagnosis or treatment for body dysmorphic disorder, disordered eating, anorexia, bulimia or clinical depression
* Pregnant

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 98 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
State Body Satisfaction | Through study completion (1 day with pretest and posttest measures)
  State body satisfaction will be measured using Visual Analogue Scales. Subjects will be asked to indicate their responses by marking a position on the scale between '0' to '100'. The three body satisfaction scales will be: 'At this moment, I am satisfied with my weight,' 'At this moment, I am satisfied with my overall appearance,' and 'At this moment, I am satisfied with my body shape.' A series of statements related to lifestyle satisfaction (i.e. relationship satisfaction, household living satisfaction, fiscal satisfaction) will also be added to this scale to uphold the cover story of this study being the effects of social media on Lifestyle Satisfaction.
State Body Appreciation | Through study completion (1 day with pretest and posttest measures)
  State body appreciation will be measured using three Visual Analogue Scales. These questions were adapted from the Body Appreciation Scale (Avalos, Tylka, & Wood-Barcalow, 2005) into state measures and were found to have high internal reliability within the previous study (Slater, Varsani, & Diedrichs, 2017). Subjects will be asked to indicate their responses by marking a position on the scale between '0' to '100'. The three body satisfaction scales will be: 'Right now, despite my flaws, I accept my body for what it is' 'right now, my feelings towards my body are positive for the most part,' and 'right now, my self-worth is independent of my body weight or shape'
State Mood | Through study completion (1 day with pretest and posttest measures)
  Subjective mood will be measured at both pre-intervention and post-intervention in the laboratory using Visual Analogue Scales. These scales will ask participants to indicate how they feel "at this moment" with regards to the following emotions: anxiety, anger, confidence, happiness, and depression

SECONDARY OUTCOMES:
Trait thin-ideal internalization | Through study completion (1 day with baseline measures only)
  Will be measured pre-exposure to the intervention images. The Sociocultural Attitudes Towards Appearance Questionnaire-4 will be included to assess this measure as an effect modifier at baseline.
Trait Social Coparison | Through study completion (1 day with baseline measures only)
  Will be measured pre-exposure to the intervention images. The Physical Appearance Comparison Scale-Revised (PACS-R) will be included to assess this measure as an effect modifier at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Der Ananian, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States